CLINICAL TRIAL: NCT00605267
Title: Multi-centre, Randomised, Double-blind, Parallel-group Study to Compare Efficacy and Safety Between Anastrozole (ZD1033) and Tamoxifen in Pre- and Post-operative Administration Under Goserelin Acetate Treatment for Premenopausal Breast Cancer Patients
Brief Title: Arimidex/Tamoxifen Neo Adjuvant Study in Premenopausal Patients With Breast Cancer Under Anti Hormonal Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D539BC00001
Record Dates: First submitted 2008-01-09; First posted 2008-01-31 (Estimated); Results first posted 2012-09-06 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2012-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Breast Neoplasms; Tumors or cancer of the human BREAST; Tumor or cancer of the human MAMMARY GLAND
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Tamoxifen; Anastrozole; Goserelin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- 1 (Active Comparator): Tamoxifen
  Interventions: Drug: Tamoxifen; Drug: Goserelin acetate (Zoladex)
- 2 (Experimental): Anastrazole (Arimidex)
  Interventions: Drug: Anastrazole (Arimidex); Drug: Goserelin acetate (Zoladex)

INTERVENTIONS:
Drug: Tamoxifen — 20 mg once daily oral dose
  Other Names: NOLVADEX
  Arms: 1
Drug: Anastrazole (Arimidex) — 1 mg once daily oral dose
  Other Names: ARIMIDEX; ZD1033
  Arms: 2
Drug: Goserelin acetate (Zoladex) — 3.6mg/month depot injection
  Other Names: ZOLADEX

SUMMARY:
The purpose of this multi-centre, randomised, double-blind, parallel-group study is to compare efficacy and safety between anastrozole and tamoxifen in pre- and post-operative administration under goserelin acetate treatment for premenopausal breast cancer patients

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal, estrogen receptor positive women, aged 20 years and over, with operable and measurable breast cancer who have provided written informed consent

Exclusion Criteria:

* Medical history of chemotherapy or endocrine therapy for breast cancer, or with treatment history of radiotherapy. Unwillingness to stop taking any drug known to affect sex hormone status (including hormone replacement therapy (HRT).

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2007-10; Primary Completion 2009-11 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Toshiyuki Kihara, Study Director — Clinical
Locations (4):
- Japan (4):
  - Research Site, Hakata, Fukuoka
  - Research Site, Kumamoto, Kumamoto
  - Research Site, Nagoya, Nagoya
  - Research Site, Osaka, Osaka

REFERENCES:
- [Derived] Masuda N, Sagara Y, Kinoshita T, Iwata H, Nakamura S, Yanagita Y, Nishimura R, Iwase H, Kamigaki S, Takei H, Noguchi S. Neoadjuvant anastrozole versus tamoxifen in patients receiving goserelin for premenopausal breast cancer (STAGE): a double-blind, randomised phase 3 trial. Lancet Oncol. 2012 Apr;13(4):345-52. doi: 10.1016/S1470-2045(11)70373-4. Epub 2012 Jan 20. PMID 22265697

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 4 research sites in Japan: Hakata (Fukuoka), Kumamoto (Kumamoto), Nagoya (Nagoya), Osaka (Osaka). The study initiation date was October 2007 and the study completion date was January 2010.
Pre-assignment Details: A total of 197 participants were recruited into this study and 98 were randomized to Anastrozole (20 mg once daily oral dose) and 99 were randomized to Tamoxifen (1 mg once daily oral dose) with one subject voluntarily discontinuing prior to receiving treatment Tamoxifen.
Groups:
- Anastrozole 1 mg: Anastrozole (investigational product) 1mg tablet given once a day orally and goserelin acetate 3.6 mg/ month depot injection
- Tamoxifen 20 mg: Tamoxifen (comparator) 20mg tablet given once a day orally and goserelin acetate 3.6 mg/ month depot injection
Period: Overall Study
Arm/Group | Anastrozole 1 mg | Tamoxifen 20 mg
Started | 98 | 99
Completed | 95 (Breast surgery performed) | 90 (Breast surgery performed)
Not Completed | 3 | 9
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 1 | 5
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anastrozole 1 mg | Tamoxifen 20 mg | Total
Number analyzed (Participants) | 98 | 99 | 197
Age, Customized [Number; unit: Participants]
  20-29 years | 2 | 0 | 2
  30-39 years | 21 | 20 | 41
  40-49 years | 65 | 68 | 133
  50-59 years | 10 | 11 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 99 | 197
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rate (BORR) (Calliper)
Description: The BORR were defined as the percentage of patients with confirmed CR or PR in the ITT population during 24 weeks pre-operative treatment period (based on the data from calliper measurement).
  CR (or PR) criteria are met at 2 or more time in points every 4 weeks. Per RECIST Criteria (V1.0) and assessed by Calliper: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >= 30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 24 weeks
Population: The BORR were defined as the percentage of patients with confirmed CR or PR in the ITT population during 24 weeks pre-operative treatment period.
  At least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter
Measure: Number; unit: Percentage of Participants
Arm/Group | Anastrozole 1 mg | Tamoxifen 20 mg
Number analyzed (Participants) | 98 | 99
Percentage of Participants | 70.4 | 50.5

2. Primary Outcome: Best Overall Response Rate (BORR) (US)
Description: The BORR were defined as the percentage of patients with confirmed CR or PR in the ITT population during 24 weeks pre-operative treatment period (based on the data from ultra sound (US) measurement).
  CR (or PR) criteria are met at 2 or more time in points every 4 weeks. Per RECIST Criteria (V1.0) and assessed by US: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >= 30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 24 weeks
Measure: Number; unit: Participants
Arm/Group | Anastrozole 1 mg | Tamoxifen 20 mg
Number analyzed (Participants) | 98 | 99
Participants | 58.2 | 42.4

3. Primary Outcome: Best Overall Response Rate (BORR) (MRI/CT)
Description: The BORR were defined as the percentage of patients with confirmed CR or PR in the ITT population during 24 weeks pre-operative treatment period(based on the data from magnetic resonance imaging (MRI) or computed tomography (CT) measurement).
  CR (or PR) criteria are met at either 12 weeks or 24 weeks. Per RECIST Criteria (V1.0) and assessed by MRI or CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >= 30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 24 weeks
Measure: Number; unit: Percentage of Participants
Arm/Group | Anastrozole 1 mg | Tamoxifen 20 mg
Number analyzed (Participants) | 98 | 99
Percentage of Participants | 64.3 | 37.4

4. Secondary Outcome: Bone Mineral Density (BMD) Lumbar Spine
Description: Change from baseline in Bone Mineral Density value (percentage), in all subjects who used DXA(Dual-energy X-ray absorptiometry) method throughout the study, at 24 weeks measured at lumbar spine.
Time Frame: Assessed at baseline and after 24 weeks of treatment
Population: The standard BMD value is defined by Japanese Osteoporosis Society in the table of reference values showing the mean for the age, gender, race, skeletal site, and densitometer measurement units was used. Then the formula was used at each measurement data: BMD(%) = Patient's BMD / standard BMD) x 100
Measure: Mean (Standard Deviation); unit: PercentageBMD=Patient's BMD/standard BMD
Arm/Group | Anastrozole 1 mg | Tamoxifen 20 mg
Number analyzed (Participants) | 80 | 78
PercentageBMD=Patient's BMD/standard BMD | -5.8 (3.4) | -2.9 (2.5)

5. Secondary Outcome: Bone Mineral Density (BMD) Cervical Thighbone
Description: Change from baseline in Bone Mineral Density value (percentage), in all subjects who used DXA(Dual-energy X-ray absorptiometry) method throughout the study, at 24 weeks measured at cervical thighbone.
Time Frame: Assessed at baseline and after 24 weeks of treatment
Population: Difference of percentage Bone Mineral Density (BMD) Cervical Thighbone = BMD percentage at 24 weeks - BMD percentage at baseline
Measure: Mean (Standard Deviation); unit: PercentageBMD=Patient'sBMD/standard BMD)
Arm/Group | Anastrozole 1 mg | Tamoxifen 20 mg
Number analyzed (Participants) | 80 | 77
PercentageBMD=Patient'sBMD/standard BMD) | -2.5 (5.1) | -0.5 (3.2)

6. Secondary Outcome: Bone Turnover Marker (BAP) EIA Method
Description: Change from baseline in serum Bone-Alkaline Phosphatase (BAP) at 24 weeks measured by EIA method
Time Frame: Assessed at baseline and after 24 weeks of treatment
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Anastrozole 1 mg | Tamoxifen 20 mg
Number analyzed (Participants) | 59 | 60
U/L | 7.1941 (6.1600) | 0.7333 (3.3640)

7. Secondary Outcome: Bone Turnover Marker (BAP) CLEIA Method
Description: Change from baseline in serum Bone-Alkaline Phosphatase (BAP) at 24 weeks measured by CLEIA method
Time Frame: Assessed at baseline and after 24 weeks of treatment
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Anastrozole 1 mg | Tamoxifen 20 mg
Number analyzed (Participants) | 36 | 30
ug/L | 3.96 (4.60) | -0.75 (3.10)

8. Secondary Outcome: Bone Turnover Marker (NTX)
Description: Change from baseline in serum crosslinked N-Telopeptide of type I collagen (NTX) at 24 weeks
Time Frame: Assessed at baseline and after 24 weeks of treatment
Measure: Mean (Standard Deviation); unit: nmolBCE(Bone Collagen Equivalent) /L
Arm/Group | Anastrozole 1 mg | Tamoxifen 20 mg
Number analyzed (Participants) | 95 | 89
nmolBCE(Bone Collagen Equivalent) /L | 9.17 (4.74) | 2.59 (3.23)

9. Secondary Outcome: Serum Oestrone (E1) Concentrations
Description: Ratio of serum Oestrone (E1) concentration (pg/mL) in the ITT population from baseline at 24 weeks.
Time Frame: Assessed at baseline and after 24 weeks of treatment
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Anastrozole 1 mg | Tamoxifen 20 mg
Number analyzed (Participants) | 96 | 92
Ratio | 0.028 (0.036) | 0.341 (0.282)

10. Secondary Outcome: Serum Oestradiol (E2) Concentrations
Description: Ratio of serum Oestradiol (E2) concentration (pg/mL) in the ITT population from baseline at 24 weeks.
Time Frame: Assessed at baseline and after 24 weeks of treatment
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Anastrozole 1 mg | Tamoxifen 20 mg
Number analyzed (Participants) | 96 | 92
Ratio | 0.041 (0.092) | 0.082 (0.186)

11. Secondary Outcome: Oestrogen Receptor (ER) Status
Description: ER status in the ITT population is categorized as Positive or Negative
Time Frame: Assessed at baseline and after 24 weeks of treatment
Measure: Number; unit: Participants
Arm/Group | Anastrozole 1 mg | Tamoxifen 20 mg
Number analyzed (Participants) | 94 | 90
Participants
  Baseline Positive & 24 weeks Negative | 2 | 1
  Baseline Positive & 24 weeks Positive | 92 | 89
  Baseline Negative & 24 weeks Negative | 0 | 0
  Baseline Negative & 24 weeks Positive | 0 | 0

12. Secondary Outcome: Progesterone Receptor (PgR) Status
Description: PgR status in the ITT population is categorized as Positive or Negative.
Time Frame: Assessed at baseline and after 24 weeks of treatment
Measure: Number; unit: Participants
Arm/Group | Anastrozole 1 mg | Tamoxifen 20 mg
Number analyzed (Participants) | 94 | 90
Participants
  Baseline Positive & 24 weeks Negative | 60 | 19
  Baseline Positive & 24 weeks Positive | 29 | 59
  Baseline Negative & 24 weeks Negative | 4 | 9
  Baseline Negative & 24 weeks Positive | 1 | 3

13. Secondary Outcome: Human Epidermal Growth Factor Receptor 2 (HER2) Status
Description: HER2 status in the ITT population is categorized as Positive or Negative
Time Frame: Assessed at baseline and after 24 weeks of treatment
Measure: Number; unit: Participants
Arm/Group | Anastrozole 1 mg | Tamoxifen 20 mg
Number analyzed (Participants) | 94 | 90
Participants
  Baseline Positive & 24 weeks Negative | 0 | 0
  Baseline Positive & 24 weeks Positive | 0 | 0
  Baseline Negative & 24 weeks Negative | 92 | 88
  Baseline Negative & 24 weeks Positive | 2 | 2

14. Secondary Outcome: Histopathological Response Rate (HRR)
Description: Number of patients in the ITT population defined as histopathological responders over the total number of patients x 100. An histopathological responder = a patient classified as Grade 1b, 2 or 3 for the histopathological response (Grade 0 = no response, 1a = mild response, 1b = moderate response, 2 = marked response or 3 = complete response)
Time Frame: Assessed at baseline and after 24 weeks of treatment
Measure: Number; unit: Percentage of Participants
Arm/Group | Anastrozole 1 mg | Tamoxifen 20 mg
Number analyzed (Participants) | 98 | 99
Percentage of Participants | 41.8 | 27.3

15. Secondary Outcome: Functional Assessment of Cancer Therapy-Breast (FACT-B)
Description: Change from baseline in Functional Assessment of Cancer Therapy-Breast (FACT-B)in the ITT population at 24 weeks. Trial Outcome Index (TOI) = the sum of the Physical Well-Being (PWB), Functional Well-Being (FWB), and Breast Cancer Scale (BCS) subscales of FACT-B.
  FACT-B includes 36 questions; 7 in PWB (Physical Well-Being); 7 inSWB (Social / Family Well-Being); 6 in EWB (Emotional Well-Being); 7 in FWB (Functional Well-Being); 9 in BCS (Breast Cancer Subscale).
  Total score of subscores or TOI is calculated from each score of question. Higher score means better and lower score means worthier.
  Score range; 0-28 in PWB; 0-28 in SWB; 0-24 in EWB; 0-28 in FWB; 0-36 in BCS; 0-92 in TOI.
Time Frame: Assessed at baseline and after 24 weeks of treatment
Population: Total score of subscores or TOI is calculated from each score of question. Higher score means better and lower score means worthier.
  PWB, FWB and BCS were assessed in this study. TOI was a total of PWB, FWB and BCS.
Measure: Mean (Standard Deviation); unit: Trial Outcome Index (TOI) (Prorated)
Arm/Group | Anastrozole 1 mg | Tamoxifen 20 mg
Number analyzed (Participants) | 95 | 92
Trial Outcome Index (TOI) (Prorated) | -4.42 (11.07) | -2.65 (8.09)

16. Secondary Outcome: Endocrine Subscale (ES)
Description: Change from baseline in Endocrine Symptom Subscale (ES)) in the ITT population at 24 weeks. ES score = the sum of the responses to all the questions on ES, low scores reflect poor quality of life and high scores reflects better quality of life.
  Score range: 0-72
Time Frame: Assessed at baseline and after 24 weeks of treatment
Population: Difference of Endocrine Subscale (ES) = ES at 24 weeks - ES at baseline.
Measure: Mean (Standard Deviation); unit: ES score
Arm/Group | Anastrozole 1 mg | Tamoxifen 20 mg
Number analyzed (Participants) | 92 | 91
ES score | -8.85 (8.69) | -6.27 (8.93)

17. Secondary Outcome: Anastrozole Plasma Concentrations (Cmin)
Description: Trough Plasma concentrations (Cmin) of Anastrozole - only Anastrozole arm was evaluated for Trough Plasma concentrations.
Time Frame: Assessed at week 12
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | Anastrozole 1 mg | Tamoxifen 20 mg
Number analyzed (Participants) | 28 | 0
ng/mL | 29.7 [17.3 to 52.4] |

ADVERSE EVENTS:
Description: One subject voluntarily discontinued prior to receiving treatment to Tamoxifen
Arm/Group | Anastrozole 1 mg | Tamoxifen 20 mg
Serious Adverse Events (participants affected / at risk) | 1/98 | 0/98
Other Adverse Events (participants affected / at risk) | 87/98 | 84/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anastrozole 1 mg (N=98) | Tamoxifen 20 mg (N=98)
Benign Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Anastrozole 1 mg (N=98) | Tamoxifen 20 mg (N=98)
Constipation (Gastrointestinal disorders) | 4 | 13
Abdominal Pain Upper (Gastrointestinal disorders) | 5 | 6
Fatigue (General disorders) | 4 | 5
Nasopharyngitis (Infections and infestations) | 27 | 24
Arthralgia (Musculoskeletal and connective tissue disorders) | 35 | 20
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 21 | 9
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 5 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 1
Headache (Nervous system disorders) | 20 | 15
Dizziness (Nervous system disorders) | 3 | 5
Hypoaesthesia (Nervous system disorders) | 5 | 3
Insomnia (Psychiatric disorders) | 7 | 9
Menopausal Symptoms (Reproductive system and breast disorders) | 6 | 4
Metrorrhagia (Reproductive system and breast disorders) | 5 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 8
Rash (Skin and subcutaneous tissue disorders) | 5 | 3
Hot Flush (Vascular disorders) | 51 | 52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less